CLINICAL TRIAL: NCT03309371
Title: DISCOGEL ®: Evaluation of the Procedure DISCOGEL ® in Lumbar Radiculopathy on Slipped Disc
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DISCOGEL
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2017-10

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lumbar disc herniation is the most important and frequent affection in rheumatology. The first treatment is based on an non-steroidal anti-inflammatory drugs.Physiotherapy also is used.But when there is no efficient result, it's usual to propose to the patient corticoid injection, percutaneous intervention or arthrodesis.

Recently DISCOGEL® is a medical device used for lumbar disc herniation. However there is no studies evaluating the benefit and the efficiency of this technic. Since a few years, the rheumatology service of GHPSJ practise this technic using DISCOGEL® with patient resistant to the medical treatment . So the aim is to evaluate the benefit of DISCOGEL® retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* age> 18
* lumbar radiculalgy
* lumbar disc herniation described by MRI
* more than 6 weeks
* prescription of DISCOGEL

Exclusion Criteria:

* medical history of surgery at the same stage
* patient under Clopidogrel or prasugrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient with a DISCOGEL treatment between January 2014 and may of 2016
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Visual Analog Scale at 2 years | Baseline, 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France